CLINICAL TRIAL: NCT04997993
Title: A Phase IA/IB Trial of Leflunomide in Patients With PTEN-Altered Advanced Solid Malignancies and HER2 Negative Breast Cancer
Brief Title: Leflunomide in Patients With PTEN-Altered Advanced Solid Malignancies and HER2 Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Deborah Doroshow (Other)
Responsible Party: Sponsor-Investigator, Deborah Doroshow, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 20-2528
Record Dates: First submitted 2021-08-02; First posted 2021-08-10 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: PTEN-Altered Advanced Solid Tumors and HER2 Negative Breast Cancer
MeSH Terms: interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Leflunomide (Experimental): Leflunomide, 20-50mg PO daily
  Interventions: Drug: Leflunomide

INTERVENTIONS:
Drug: Leflunomide — Leflunomide, 20-50mg PO daily

SUMMARY:
Leflunomide in patients with PTEN-Altered advanced solid tumors or HER2 negative breast cancer. Phase 1A objectives are to determine the safety, tolerability, and the MTD of leflunomide in patients with PTEN-Altered advanced solid malignancies and HER2 negative breast cancer. Phase 1B objective is to assess preliminary evidence of clinical activity of leflunomide in these patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* A) Advanced or metastatic solid tumor with lack of PTEN expression as determined by immunohistochemistry. Lack of PTEN expression is defined as the absence of staining in the tumor (<5%), with strong positive staining of adjacent normal endometrium or stromal cells, using the monoclonal DAKO antibody 6H2.1.9 OR
* B) Advanced or metastatic solid tumor with a deleterious somatic mutation in PTEN as determined by tissue or ctDNA testing in a CLIA laboratory and classified as deleterious in the ClinVar or COSMIC databases OR
* C) Advanced or metastatic HER2 negative breast cancer. Patients must have received ≤ 3 prior cytotoxic chemotherapies for metastatic disease (immunotherapy does not count as a line of therapy), and up to 2 prior antibody drug conjugate regimens (eg, sacituzumab govitecan, trastuzumab deruxtecan). Patients with ER-positive breast cancer (ER>10%) are eligible if they have had progressive disease after at least 1 prior CKD4/6 inhibitor. Patients must have received alpelisib or capivasertib if eligible for either therapy or must be intolerant to or have refused such therapy.

  °Patients with known PTEN altered breast cancer may participate regardless of lines of prior therapy if they meet criteria A or B.
* Measurable disease only required for dose expansion in non-prostate ca patients
* Patients with prostate cancer without measurable disease must have evaluable disease as assessed by serum PSA.
* Patients must have progressed on, be refractory or intolerant of standard therapy for their cancer, if such a standard therapy exists.
* Patients with treated brain metastases are eligible if follow-up brain imaging at least 4 weeks after CNS directed therapy shows no evidence of progression.
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS directed therapy is not required and is unlikely to be required during the first cycle of therapy.
* 2 week or five half life treatment (whichever is shorter) washout from systemic therapy, surgery, or RT. Patients with prostate cancer receiving gonadotropin-releasing hormone agonists may continue their use while on study.
* ECOG performance status 0-2.
* Patients with HIV on effective anti-retroviral therapy with an undetectable viral load are eligible for this trial.
* Adequate organ and marrow function as defined below:
* Leukocytes ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,000/mcL
* Platelets ≥ 100,000/mcl
* Total bilirubin ≤ 1.5 x ULN (or direct bilirubin, if patient has Gilbert's disease)
* AST (SGOT)/ALT (SPGT) ≤ 3xULN
* GFR (Cockroft-Gault) ≥ 40 mL/min/1.73m2
* Negative serum or urine pregnancy test within 3 days prior to C1D1 of leflunomide therapy.
* Women of child-bearing potential and men must agree to use adequate contraception before study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately and will immediately be taken off study therapy.
* Additionally, all women of child bearing potential must begin an accelerated elimination protocol upon drug discontinuation for any reason, unless they agree to continue taking appropriate contraception for up to 2 years from study drug discontinuation.
* Patients who do not take the accelerated elimination protocol will have to remain on contraception for two years.
* Recommended methods of birth control are: The consistent use of an approved hormonal contraception such as an intrauterine device (IUD), birth control pills, double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), sexual abstinence (no sexual intercourse) or sterilization.

A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 months).
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients with primary CNS tumors are not eligible.
* Patients who have had chemotherapy or radiotherapy within 4 weeks before entering the study or those who have not recovered from grade ≥ 2 adverse events due to agents administered more than 4 weeks earlier. Adverse events such as alopecia, hypothyroidism, and neuropathy are allowed. Other adverse events may be allowed by permission of the principal investigator.
* Patients may not be receiving any other investigational agents.
* A known history of acute or chronic Hepatitis B or C, due to the known potential hepatotoxicity of leflunomide.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to leflunomide or teriflunomide.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose-limiting toxicities | 1 month
  Grade 3 or higher non-hematologic toxicity, Any death not clearly due to the underlying disease, Cases defined by Hy's law, Grade 4 neutropenia or thrombocytopenia > 7 days, Grade 3 thrombocytopenia with clinically significant bleeding, Febrile neutropenia
Number of Dose-limiting toxicities | 1 month
  Grade 3 or higher non-hematologic toxicity Any death not clearly due to the underlying disease Cases defined by Hy's law Grade 4 neutropenia or thrombocytopenia > 7 days Grade 3 thrombocytopenia with clinically significant bleeding Febrile neutropenia

SECONDARY OUTCOMES:
Maximum tolerated dose | 2 years
  A standard 3+3 design is used to define the MTD. Dose level 0 will only be utilized in the presence of ≥2/6 DLTs in dose level 1 or for a dose reduction if a patient does not tolerate dose level one. Standard dosing for rheumatoid arthritis is 100mg daily for 3 days loading dose followed by 20mg daily maintenance dose, which can be reduced to 10mg in the event of intolerance.
Overall Response Rate | 2 years
  Overall Response Rate for dose expansion cohort. Overall response rate is defined as the proportion of patients achieving a best response of complete response or partial response using RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Doroshow, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available